CLINICAL TRIAL: NCT01659463
Title: Resin Infiltration on Teh Sealing of Proximal Early Caries Lesins: a Randomized Trial
Brief Title: Resin Infiltratration on the Sealing of Proximal Early Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Julio Eduardo do Amaral, MsC, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0347.0243.000-10
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Tooth; Lesion, White Spot Lesions
Keywords: CARIES INFILTRATION; CARIES LESION; INFILTRANT

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICON - low viscosity resin (Experimental): APPLICATION OF A LOW VISCOSITY RESIN IN EARLY PROXIMAL CARIES LESIONS
  Interventions: Other: ICON
- INSTRUCTIONS ORAL HYGIENE (Active Comparator): INSTRUCTION ORAL HYGIENE AND DIET AND TOOPICAL FLUORIDE APPLICATIONS
  Interventions: Behavioral: instruction oral hygiene

INTERVENTIONS:
Other: ICON — LOW VISCOSITY RESIN WILL BE APPLIED IN EARLY PROXIMAL CARIES LESIONS
  Other Names: ICON (DMG) Hamburg Germany
  Arms: ICON - low viscosity resin
Behavioral: instruction oral hygiene — Instructions diet and hygiene oral and topical fluoride
  Arms: INSTRUCTIONS ORAL HYGIENE

SUMMARY:
Material for caries prevention dont have better results compared with non-operatory interventions.

DETAILED DESCRIPTION:
Two gruops will be compared. One using ICON and another gruop with non-operatory interventions consisted in hygiene instrutions and fluoride topical application. The caries progression will be evalueted with radiographic observation.

ELIGIBILITY:
Inclusion Criteria:

* Two early caries lesion in the same patient, lesion with the same radiolucencies images

Exclusion Criteria:

* Pregnancy, use of orthodontics appliences, use of drugs modified salivar flow, ausence of adjacent teeth

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
caries progression in the proximal surfaces | One year after interventions
  progression in the proximal surfaces will be compared with two procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Julio E Zenkner, MsC, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil